CLINICAL TRIAL: NCT02339896
Title: Observation an Immunogenicity and Safety Study of Modified TRC-ID Regimen With A New Chromatographically Purified Vero Cell Rabies Vaccine (SPEEDA®) With or Without Rabies Immunoglobulin in Children
Brief Title: Observation Study an Immunogenicity Modified TRC-ID Regimen With CPRV With or Without Rabies Immunoglobulin in Children
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Piyada Angsuwatcharakon, MD, Queen Saovabha Memorial Institute
Other Study IDs: RC5704
Record Dates: First submitted 2015-01-07; First posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Dog Bite
Keywords: rabies; modified TRC intradermal rabies vaccine; SPEEDA
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Biospecimen Retention: Samples Without DNA — Rabies Neutralizing antibody
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- WHO category 2: Children patient who have experienced WHO category II exposure will receive rabies vaccine (SPEEDA) 0.1 ml intradermal two site for 4 times
  Interventions: Biological: rabies vaccine
- WHO category 3: Children patient who have experienced WHO category II exposure will receive rabies vaccine (SPEEDA) 0.1 ml intradermal two site for 4 times with ERIG
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: rabies vaccine — rabies vaccine 0.1 ml intradermal two site for 4 times

SUMMARY:
To determine Immunogenicity and Safety Study of Modified TRC-ID Regimen with A New Chromatographically Purified Vero Cell Rabies Vaccine (SPEEDA®) as post exposure rabies intradermal regimen with or without Rabies Immunoglobulin in Children

DETAILED DESCRIPTION:
post exposure rabies vaccination with modified Thai red cross intrademal regimen has been proven to be immunogenic and effection when using purified vero cell vaccine (PVRV) In present, new chromatographically purified vero cell rabies vaccine (SPEEDA), chromatography purifed vero cell derived rabies vaccine, is manufactured by the Liaoning Chengda Biotechnology is available This study has a goal to determine the immunogenicity of speeda when using with post exposure rabies intradermal vaccination with or without rabies immune globulin in children

ELIGIBILITY:
Inclusion Criteria:

* they are 1-15 years healthy children
* give signed informed consent from their parents
* willing to participate in this study and be able to receive the vaccination and collect blood sample as the study plan.

Exclusion Criteria:

* they have prior history of rabies vaccination or any equine/human serum administration such as snake antivenom and tetanus antiserum or vaccine allergy
* Persons who have immunosuppressive conditions such as known HIV infection, transplantation, chronic renal failure, receiving of steroid or immunosuppressive drugs
* person received anti-malarial drugs within the previous two months or any blood products within previous three months were excluded
* Urine pregnancy test must be done in all female adolescents to exclude the pregnancy in first visit

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: recruit the patients from Rabies clinic of Queen Saovabha Memorial Institute, Thammasat Hospital, Charoen Krung Pracha Rak Hospital and HRM Princess Maha Chakri Sirindhorn Medical Center and all had experienced WHO category II or III exposure to suspected rabid animal. In patients with WHO category III have to receive a heterologous biological (ERIG or HRIG)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
determine the level of rabies neutralizing antibodies after using SPEEDA® with modified TRC-ID rabies with or without RIG and the safety of using SPEEDA® with modified TRC-ID rabies with or without RIG in children | 1 year 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Piyada Angsuwatcharakon, MD, Principal Investigator — QSMI TRC society